CLINICAL TRIAL: NCT04718974
Title: Acceptability, Effect and Cost of Mobile-health on ART Adherence Among Youths: A Mixed Methods Sequential Study in Kiryandongo
Brief Title: Call for Life Youth ART Adherence Study
Acronym: C4L-Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: Infectious Diseases Institute, Uganda (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IDI-SRC Ref: 031/2019; UNCST Folio Number: HS576ES (Other: UNCST( Uganda National Council for Science & Technology)); HDREC #REC Ref: 2019-083 (Other: School of Medicine,Higher Degrees Research Ethics Committee)
Record Dates: First submitted 2021-01-06; First posted 2021-01-22 (Actual); Results first posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2023-07

CONDITIONS: ART Adherence; HIV-1-infection; mHealth
Keywords: Youth; Adherence; ART; mobile health; resource poor setting
MeSH Terms: interventions — CD56 Antigen

STUDY DESIGN:
Intervention Model Description: 2 groups one on intervention of Call for life mHealth with standard of care and other on standard of care only.
  mHealth Call for life Tool using interactive voice response
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention " Call for life- mHealth tool" with standard of care for PLHIV (Experimental): The system has options to either use interactive voice response or short message service and the user has to make a choice, get a secret pin code which ensures privacy to end user.
  The mHealth tool/system offers personalised pill reminder calls, health tip messages, clinic appointment reminders and remote symptom reporting
  Interventions: Other: mHealth call for life system/ tool using IVR ( interactive voice response)
- Standard of care "usual care" (No Intervention): Standard
  • Care and support for people living with HIV, and the first line ART regimen is based on the Apr 2018, consolidated guidelines for prevention and treatment of HIV in Uganda (MoH, 2018), and will also follow the healthcare services package for PLHIV including the Adult Care and Treatment Package.

INTERVENTIONS:
Other: mHealth call for life system/ tool using IVR ( interactive voice response) — The tool capitalises on a basic mobile phone's core utilities of voice and short messaging services. The system design, development, testing and evaluation was done by Janssen and the Grameen Foundation (http://motechsuite.org/index.php/implementations). In 2015, Janssen Global Public Health Research and Development, in close collaboration with the Infectious Diseases Institute Kampala (IDI), developed Call for Life Uganda (CFLU) tailored to the needs of PLHIV in Uganda
  Other Names: Call for life -mHealth tool
  Arms: intervention " Call for life- mHealth tool" with standard of care for PLHIV

SUMMARY:
Study purpose: To assess effect of mHealth Call for life Uganda tool (CFLU) on ART adherence among youth measured by interactive voice response to daily adherence calls mapped in the database and proportion with viral suppression of copies below 1000 copies/mL.

The intervention call for life Uganda (CFLU) uses IVR calls or text messages delivered via MOTECH™ based Connect for Life technology™. The calls are delivered in 4 languages (Luganda, English, Luo and Runyakitara) and the participant has to make a choice of the preferred language during registration to the system. The system offers adherence pill reminders, health message tips, visit appointment reminders and receipt of self-reported symptoms.

DETAILED DESCRIPTION:
The intervention is mobile phone based IVR. However, the CLFU trial found that, it was observed that a good number of participants (50 of 256) at the urban site were not enrolled due to absence of a basic mobile phone, or had malfunctioning phone keyboards (for Poster Exhibition at the 20th International Conference on AIDS and STIs in Africa (ICASA 2019). Therefore, we shall provide a basic mobile phone to everyone in the study (SoC and intervention arm). To avoid stigma associated with a particular phone, we shall get 4 or more types of basic phones. Issues regarding simcard registration will be dealt with by the individuals.

Four study questionnaires will be administered at baseline and 6-monthly until the 12-month exit visit.

The questionnaires will capture:

* Sociodemographic and medical history
* Stigma scores
* Knowledge assessment
* Sexual behavior assessment
* Knowledge of COVID-19 ( only at baseline) The data will be entered using REDCap. Blood for viral load will be collected at baseline and at the 6 and 12-month visit.

Intervention: mHealth CFLU tool The tool capitalises on a basic mobile phone's core utilities of voice and short messaging services. The system design, development, testing and evaluation was done by Janssen and the Grameen Foundation (http://motechsuite.org/index.php/implementations). In 2015, Janssen Global Public Health Research and Development, in close collaboration with the Infectious Diseases Institute Kampala (IDI), developed Call for Life Uganda (CFLU) tailored to the needs of PLHIV in Uganda. The CFLU system follows the Health Insurance Portability and Accountability Act (HIPAA) Privacy and Security rules. While the Privacy rules deals with electronic Protected Health Information, the security rule covers administrative, physical and technical safeguards to ensure confidentiality, integrity and security of electronic protected health information. Data transaction between patient and system is encrypted when it comes to human subjects. The system is password protected, and interaction of system and patient is personalised with a secret code. The system interacts with the patient through a basic mobile phone via a keypad and with the health worker through a web-based interface. The system has options to either use interactive voice response or short message service and the user has to make a choice, get a secret pin code which ensures privacy to enduser.

Screening-Enrolment procedures:

All potential participants will be written on the screening log, and a screening form completed, reasons for screen failure will be documented on the screening log. Following successful screening, the participant will be referred to the Research Assistant (RA) to receive a thorough explanation of the study so and informed consent is obtained. The RA then administers the stigma questionnaire along with the sociodemographic and medical information, , HIV knowledge and sexual behaviour questionnaires. A client locater form will be completed which will help in physical contact tracing, and the participant will be registered on the enrolment log.

Randomisation will follow (see details of randomisation procedure below) thereafter and the result in the sealed envelope will dictate whether the patient will be registered onto the Call for Life System for the intervention or continue with standard of care as per Ministry of Health HIV Management guidelines.

Registration onto the CFLU system: Refer to Standard operating procedures on registration.

However, all patients will be registered onto the electronic and hard copy of the enrolment log and a next appointment date is given to them. Finally, the lab request forms are filled and the patient sent for a blood draw. The patient returns from the lab, receives their transport refund of UGX 20,000, with a basic mobile phone (only at baseline visit, to all participants) and is allowed to go home.

No intervention: Standard of care arm The Ministry of Health developed a minimum healthcare services package for PLHIV to standardize the programming, implementation and delivery of integrated HIV services in Uganda The standard of care arm is based on the Apr 2018, consolidated guidelines for prevention and treatment of HIV in Uganda (MoH, 2018), and will also follow the healthcare services package for PLHIV (Uganda. MoH, September 2014).

ELIGIBILITY:
Inclusion Criteria:

* Youth living with HIV
* Documented HIV test result
* ART naïve or on ART since Jun 2019

Exclusion Criteria:

* Youth with Hearing loss,
* Youth with severe illness likely to shorten life span,
* Youth in boarding schools
* Inability to use a basic mobile phone

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 206 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Agnes B Naggirinya, MMed, Principal Investigator — Infectious Diseases Institute
Locations (1):
- Kiryandongo, Kiryandongo, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bwanika Naggirinya A, Meya DB, Nabaggala MS, Banturaki G, Kiragga A, Rujumba J, Waiswa P, Parkes-Ratanshi R. Effectiveness of interactive voice response-call for life mHealth tool on adherence to anti-retroviral therapy among young people living with HIV: A randomized trial in Uganda. PLoS One. 2024 Nov 19;19(11):e0308923. doi: 10.1371/journal.pone.0308923. eCollection 2024. PMID 39561129

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started on 12th Aug 2020. Reccruitment was from three HIV/ART clinics in Kiryandongo District
Pre-assignment Details: The participants must have registered in either of the three study site. They should have been between 15-24 years and on ART for 6 months or less.
Groups:
- Intervention " Call for Life- mHealth Tool" With Standard of Care for PLHIV: The system has options to either use interactive voice response or short message service and the user has to make a choice, get a secret pin code which ensures privacy to end user.
  The mHealth tool/system offers personalised pill reminder calls, health tip messages, clinic appointment reminders and remote symptom reporting
  mHealth call for life system/ tool using IVR ( interactive voice response): The tool capitalises on a basic mobile phone's core utilities of voice and short messaging services. The system design, development, testing and evaluation was done by Janssen and the Grameen Foundation (http://motechsuite.org/index.php/implementations). In 2015, Janssen Global Public Health Research and Development, in close collaboration with the Infectious Diseases Institute Kampala (IDI), developed Call for Life Uganda (CFLU) tailored to the needs of PLHIV in Uganda
Period: Overall Study
Arm/Group | Intervention " Call for Life- mHealth Tool" With Standard of Care for PLHIV | Standard of Care "Usual Care"
Started | 103 (We started with 103 participants, at baseline, they were provided with a basic cellphone, were registered on the intervention which offered individualised daily pill reminders, clinic appointment reminders, weekly voice health information and remote symptom management via toll free number to call in whenever in need. In addition,participants received the standard of care which includes facility based counselling, ART counseling and facility based health education talks at pill refills.) | 103 (Participants received services based on standard of care per Ministry of Health guidelines, not limited to; facility based counselling,pill refills based on duration on ART with those initiating having frequent visits, ART counselling, facility based health education talks. They were seen every 6 months until 12 months as per protocol.)
Completed | 91 (Number of participants that turned up for month 12 follow-up were 91) | 77 (Number of participants that turned up at month 12 follow-up were 77)
Not Completed | 12 | 26
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 10 | 20
Not completed — Transferred out | 2 | 4

BASELINE CHARACTERISTICS:
Population: Young people 15-24 years initiating or on ART since 2019.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention " Call for Life- mHealth Tool" With Standard of Care for PLHIV | Standard of Care "Usual Care" | Total
Number analyzed (Participants) | 103 | 103 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.5 (1.9) | 22.2 (2.3) | 22.3 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 85 | 167
  Male | 21 | 18 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — All participants were from the Black African Race
  Participants
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 0 | 0 | 0
    Unknown or Not Reported | 103 | 103 | 206
Region of Enrollment [Count of Participants; unit: Participants] — All participants were recruited from Kiryandongo district, North-Western Uganda region
  Participants
    Uganda | 103 | 103 | 206
Viral load detection at baseline [Count of Participants; unit: Participants] | 46 | 32 | 78

OUTCOME MEASURES:

1. Primary Outcome: • Viral Load Suppression
Description: Viral load suppression as per Blood draws at 6 months for those on intervention and those on standard of care arm will be used to measure viral load at these time points
Time Frame: • Viral load suppression at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention " Call for Life- mHealth Tool" With Standard of Care for PLHIV | Standard of Care "Usual Care"
Number analyzed (Participants) | 96 | 87
Participants | 61 | 46

2. Primary Outcome: • Viral Load Suppression
Description: Viral load suppression as per Blood draws at 12 months for those on intervention and those on standard of care arm will be used to measure viral load status at these time points
Time Frame: • Viral load suppression at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention " Call for Life- mHealth Tool" With Standard of Care for PLHIV | Standard of Care "Usual Care"
Number analyzed (Participants) | 91 | 77
Participants | 67 | 40

3. Primary Outcome: Proportions Retained in Care
Description: Proportions of youth retained in care at 12 months for those on intervention in comparison to those on standard of care arm
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention " Call for Life- mHealth Tool" With Standard of Care for PLHIV | Standard of Care "Usual Care"
Number analyzed (Participants) | 103 | 103
Participants | 91 | 77

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from participant randomization until exit. This period was 1year and 9 months.
Description: ICH E6 Section 1.2. 5. • An adverse event can be any unfavorable and unintended sign, symptom, or disease that occurs to a study participant, even if not related to the intervention under study.
  An AE becomes serious if it results into: Death. A life-threatening adverse event. Inpatient hospitalization, or prolonged of existing hospitalization. A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions. A congenital anomaly/birth defect.
Arm/Group | Intervention " Call for Life- mHealth Tool" With Standard of Care for PLHIV | Standard of Care "Usual Care"
All-Cause Mortality (participants affected / at risk) | 0/103 | 2/103
Serious Adverse Events (participants affected / at risk) | 1/103 | 2/103
Other Adverse Events (participants affected / at risk) | 0/103 | 0/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention " Call for Life- mHealth Tool" With Standard of Care for PLHIV (N=103) | Standard of Care "Usual Care" (N=103)
Death (Infections and infestations) | 0 (0) | 2 (2)
Road traffic Accident (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Participant was knocked while riding on a motorcycle

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/74/NCT04718974/Prot_SAP_ICF_000.pdf